CLINICAL TRIAL: NCT01892462
Title: Circulating Biomarkers and Ventricular Tachyarrhythmia
Acronym: LIFEMARKER
Status: Completed | Type: Observational
Sponsor: Ochsner Health System (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Daniel P Morin, MD MPH FHRS, Cardiac Electrophysiologist, Director of Cardiovascular Research, Ochsner Health System
Other Study IDs: ISRCRM400003
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Cardiomyopathy; Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Cardiomyopathies; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be stored frozen for future analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether levels of inflammatory markers in circulating blood can correlate with risk for dangerous heart rhythms. Patients with systolic heart failure, which has been shown to increase risk for dangerous heart rhythms, will be enrolled. All subjects will have an implantable cardioverter-defibrillator (ICD) in place, which allows regular evaluation of heart rhythm.

DETAILED DESCRIPTION:
If you agree to be in this study, you will be asked to the following things:

* you will come into the EP device clinic every three months for one year to have your device interrogated and will complete an EKG
* you will have labs drawn to measure levels of certain markers of inflammation in the body. This information will be used to identify new ways to test for risk of abnormal heart rhythms and other heart disease
* you will review your medications with the study coordinator and along with any recent illnesses or hospitalizations

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction [LVEF] <=35%
* ICD implant

Exclusion Criteria:

* Recent myocardial infarction (12 weeks)
* Recent revascularization (12 weeks)
* Recent hospitalization for any cause (6 weeks)
* History of rheumatologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiomyopathy (left ventricular ejection fraction [LVEF] <=35%) who are followed at our institution's ICD device clinic will have levels of circulating biomarkers (hs-CRP, IL-6, TNF-alpha, IL-1, sST2, MMP-1, CICP, CITP) and BNP assessed at three-month intervals for at least one year. Patients will be excluded from the study if they have had a recent myocardial infarction or PCI (within three months), or recent hospitalization.
  Patients with obvious primary inflammatory conditions (such as lupus and rheumatoid arthritis) will be excluded. Additionally, significant events (e.g., HF hospitalizations, revascularization, medication changes, and death) will be tracked at each follow up visit for further statistical analysis.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
to evaluate a large population of heart failure patients with regard to circulating biomarkers and rates of subsequent ventricular arrhythmias. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Morin, MD MPH, Principal Investigator — Ochsner Medical Foundation
Locations (1):
- Ochsner Health System, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Morin DP, Chong-Yik R, Thihalolipavan S, Krauthammer YS, Bernard ML, Khatib S, Polin GM, Rogers PA. Utility of serial measurement of biomarkers of cardiovascular stress and inflammation in systolic dysfunction. Europace. 2020 Jul 1;22(7):1044-1053. doi: 10.1093/europace/euaa075. PMID 32357207